CLINICAL TRIAL: NCT06050083
Title: Digital Clinical Hypnosis for Chronic Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor: School of Medicine Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014786; R41AT011996 (NIH)
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain; Chronic Pain
Keywords: Low-back Pain; Hypnosis; Chronic Pain; Digital Health
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Study 1 and 2 are both 2-arm randomized controlled trials in which individuals are randomly assigned to a treatment group (8 weeks of access to hypnosis recordings) or a waitlist group (4 weeks of no access followed by 4 weeks of access to hypnosis recording access).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 8 weeks of access to Rose web application (online hypnosis recordings)
  Interventions: Behavioral: Hypnosis audio recordings
- Waitlist Control (Active Comparator): 4 weeks of waitlist (no access to Rose application for 4 weeks and then 4 weeks of access to Rose web application)
  Interventions: Behavioral: Hypnosis audio recordings

INTERVENTIONS:
Behavioral: Hypnosis audio recordings — A web application (Rose) that contains hypnosis audio recordings created by the investigators.

SUMMARY:
This ClinicalTrials.gov posting contains two randomized controlled trials. The study procedures were identical, except Study 1 was funded by NIH and enrolled adults with chronic low back pain, whereas Study 2 was funded by the UW Department of Rehabilitation Medicine and enrolled adults with any type of chronic pain. Study 1 and 2 each enrolled 50 adults (N = 100 total across the two studies). Although Study 2 did not use NIH funds, we are including the results here because the studies were conducted simultaneously by the same PI (Dr. Jensen) with the same study procedures.

Participants enrolled in the studies for a duration of 8 weeks. The studies test the feasibility and efficacy of a therapeutic hypnosis digital application (website), called Rose. The investigators wanted to determine if the Rose application was user-friendly and effective at improving quality of life and reducing pain for adults with chronic pain. If successfuly, the investigators hope to develop the Rose application into a mobile app that will be publicly available and managed by HypnoScientific Inc., a company that is co-owned by the investigators.

Participants completed brief (15-20min) self-report surveys that ask about pain and mental health at three timepoints: Baseline (week 0), 4 weeks, and 8 weeks.

DETAILED DESCRIPTION:
Pain is a major public health problem that affects over 100 million adults in the United States. While pain can have profound negative impacts, current treatment remains inadequate. A focus on opioid treatments has led to over-prescription, harmful side effects, and the overuse crisis. To address this problem, the study investigators, and others, have developed and adapted hypnosis to empower individuals to self-manage pain. Findings from the investigators' research supports hypnosis as an effective non-pharmacological technique. However, a significant limitation of hypnosis treatment is access, given that hypnosis treatment is provided by a very limited number of clinicians with training in its use, as well as the significant costs of in-person treatment.

The main goal of this study is to pilot test the efficacy of hypnosis content for pain management as provided via recordings in the Rose web application.

ELIGIBILITY:
Inclusion Criteria (self-report online and telephone screening by study staff):

* 18 years old or older
* Chronic Pain or Chronic Low Back Pain (i.e., pain in the low back that has been an ongoing problem for 3 months or more for at least half the days, as disclosed during self-report screening. The pain can be a primary condition or secondary to another health condition.
* Average pain intensity in the past week ≥ 4 on a 0-10 scale
* Reads, speaks, and understands English as noted in the medical record or disclosed during self-report screening
* Has regular access to the internet
* Has access to devices (phone, desktop, or other) with features (browsers, audio capabilities, etc.) that are congruent with the requirements of the digital therapeutic, as assessed by staff members during self-report screening.

Exclusion Criteria:

* History of (within past 5 years) or current diagnosis of primary psychotic or major thought disorder with active symptoms as noted in the medical record or disclosed during self-report screening
* Psychiatric hospitalization within the past 6 months as noted in the medical record or disclosed during self-report screening
* Psychiatric or behavioral conditions in which symptoms were unstable or severe within the past 6 months as noted in the medical record or disclosed during self-report screening;
* Any psychiatric or behavioral issues as noted in the medical record or disclosed/observed during self-report screening that would indicate subject may be inappropriate for study;
* Presenting symptoms at the time of screening that would interfere with participation, specifically active suicidal ideation with intent to harm oneself or others or active delusional or psychotic thinking;
* Active malignancy (e.g., cancer not in remission) as noted in the medical record or disclosed during self-report screening;
* Pain condition for which surgery is recommended and/or planned in the next six months as disclosed during self-report screening;
* Currently receiving or have received hypnosis treatment for any pain condition as disclosed during self-report screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, School of Medicine, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primarily recruited from Research Match and the UW Rehabilitation Medicine Participant Pool.
Groups:
- Study 1: 8 Week Treatment: Participants that had access to the Rose application for 8 weeks.
- Study 1: 4 Week Waitlist; Study 2: 4 Week Waitlist: 4 Week Waitlist (4 weeks waitlist, then 4 weeks of Rose application access)
- Study 2: 8 Week Treatment: Participants had access to the Rose application for 8 weeks.
Period: Overall Study
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Started | 26 | 24 | 26 | 24
Completed | 26 | 24 | 26 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of participants per study group in Study 1 and Study 2
Groups:
- Study 1: 4 Week Waitlist; Study 2: 4 Week Waitlist: Participants that had access to the Rose application for 4 weeks (8 weeks total participation = 4 weeks waitlist with no access to the Rose application, then 4 weeks of access)
- Total: Total of all reporting groups
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist | Total
Number analyzed (Participants) | 26 | 24 | 26 | 24 | 100
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex Assigned at Birth (Female, Male)
  Participants
    Sex at Birth: Female | 19 | 18 | 12 | 12 | 61
    Sex at Birth: Male | 7 | 6 | 14 | 12 | 39
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender Identity (Female, Male, Transgender, Non-binary)
  Participants
    Gender: Female | 19 | 17 | 11 | 12 | 59
    Gender: Male | 7 | 6 | 12 | 12 | 37
    Gender: Transgender | 0 | 1 | 2 | 0 | 3
    Gender: Non-binary | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (Hispanic/Latinx or Non-Hispanic/Latinx)
  Participants
    Hispanic or Latino | 6 | 5 | 1 | 3 | 15
    Not Hispanic or Latino | 19 | 19 | 25 | 21 | 84
    Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (using NIH Racial Identity categories)
  Participants
    American Indian or Alaska Native | 2 | 1 | 0 | 0 | 3
    Asian | 1 | 1 | 1 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 9 | 7 | 15 | 13 | 44
    White | 10 | 11 | 8 | 10 | 39
    More than one race | 4 | 3 | 2 | 1 | 10
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Geographical Region of Enrollment
  Participants
    United States | 26 | 24 | 26 | 24 | 100
Years of Education [Count of Participants; unit: Participants] — Number of years of education
  Participants
    High School Graduate/GED | 2 | 2 | 1 | 1 | 6
    Some college or vocational school | 10 | 11 | 2 | 5 | 28
    2 year college graduate | 5 | 4 | 3 | 0 | 12
    4 year college graduate | 3 | 6 | 7 | 3 | 19
    Graduate school | 6 | 1 | 13 | 15 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age measured as a continuous variable
  Years | 48.3 (20.8) | 49.5 (15.6) | 38.6 (12.7) | 40.6 (16.7) | 48.9 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Using Rose Application
Description: Total # of hypnosis sessions listened to by participants
Time Frame: During the 8 weeks of study participation
Population: The number of hypnosis sessions listened to was prespecified to be aggregated for all participants because (1) it was over the entire course of the 8-week study and participants in both arms had access and (2) the key variable of interest for feasibility was any difference in the number and rate of listening as a function of session duration (and not differences as a function of condition, as those in the waitlist condition would by default listen to fewer sessions).
Measure: Number; unit: # of hypnosis sessions listened to
Groups:
- Study 1: Summary scores for all participants in both the Treatment/Control groups for Study 1.
- Study 2: Summary scores for all participants in both the Treatment/Control groups for Study 2.
Arm/Group | Study 1 | Study 2
Number analyzed (Participants) | 50 | 50
# of hypnosis sessions listened to
  5 minute audio recording | 81 | 79
  10 minute audio recording | 64 | 134
  20 minute audio recording | 220 | 274

2. Primary Outcome: Continued Interest in Using Rose Application
Description: Participants reporting how interested they would be in continuing to use the Rose application: "If the Rose web/phone application were available to download, how interested would you be in downloading and using this application?" 4 - Extremely interested 3 - Very interested 2 - Somewhat interested
  1 - Little interested 0 - Not interested
Time Frame: 8 week assessment
Population: The number of participants who expressed expressed am interest in continued interest access to the application was prespecified to be aggregated for all participants because the milestone for this feasibility variable was the overall rate of interest in for those who used the application at least once, collapsed across condition. We were not interested in, or anticipated, any between-group difference in this variable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Study 1: Overall results for Study 1
- Study 2: Overall results for Study 2
Arm/Group | Study 1 | Study 2
Number analyzed (Participants) | 50 | 50
Score on a scale | 2.5 (1.3) | 2.8 (1.5)

3. Primary Outcome: Willingness to Pay for Continued Use of Rose Application
Description: Participants that reported a willingness to pay for continued access to the Rose application (results available for Study 2 only): "Would you be willing to pay some amount for a monthly subscription to Rose, to have continued access?"
  1 - Yes 0 - No
Time Frame: 8 week assessment
Population: The number of participants who expressed a willingness to pay fo continued access to the application was prespecified to be aggregated for all participants because the milestone for this feasibility variable was the overall rate of willingness to pay for the application for those who used the application at least once, collapsed across condition. We were not interested in, or anticipated, any between-group difference in this variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 2
Number analyzed (Participants) | 17
Participants | 11

4. Secondary Outcome: Average Pain - Past Week
Description: A 0-10 Numerical Rating scale of average pain in the past week: "Please rate your pain by choosing the one number that best describes your pain at its WORST in the PAST WEEK, where 0 is "no pain" and 10 is "pain as bad as you can imagine"
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
Score on a scale
  Baseline | 5.81 (1.44) | 5.71 (1.88) | 5.92 (1.70) | 5.83 (1.83)
  4 Weeks | 5.69 (1.74) | 5.42 (1.79) | 5.04 (1.51) | 5.17 (1.49)
  8 Weeks | 5.38 (2.12) | 4.96 (1.72) | 4.46 (1.84) | 3.46 (2.08)

5. Secondary Outcome: Worst Pain - Past Week
Description: A 0-10 Numerical Rating scale of worst pain in the past week: "Please rate your pain by choosing the one number that best describes your pain at its WORST in the PAST WEEK, where 0 is "no pain" and 10 is "pain as bad as you can imagine"
Time Frame: Baseline, 4 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
Score on a scale
  Baseline | 7.23 (1.34) | 7.63 (1.38) | 7.35 (1.02) | 7.29 (0.95)
  4 Weeks | 7.19 (1.60) | 6.92 (1.47) | 6.16 (1.57) | 6.63 (1.35)
  8 Weeks | 6.69 (1.91) | 6.91 (1.81) | 5.73 (2.39) | 4.96 (2.39)

6. Secondary Outcome: PROMIS Sleep Disturbance Short Form 8a
Description: Domain assessed: Sleep Disturbance. Ratings are summed and converted to T scores (Mean = 50 and SD = 10 in the normative sample).
  Higher scores indicate more sleep disturbance. Scores that are >= 55 (i.e., one half a SD above the normative mean) are considered clinically elevated.
Time Frame: Baseline (week 0), 4 week assessment, 8 week assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
T-score
  Baseline | 57.3 (7.9) | 58.5 (8.7) | 55.2 (7.4) | 57.2 (9.5)
  4 Weeks | 58.4 (9.7) | 57.3 (9.1) | 41.7 (10.7) | 54.0 (10.2)
  8 Weeks | 57.1 (10.0) | 53.5 (10.8) | 50.5 (10.6) | 50.0 (12.6)

7. Secondary Outcome: PROMIS Pain Interference Short Form
Description: Domain assessed: Pain interference. Ratings are summed and converted to T scores (Mean = 50 and SD = 10 in the normative sample).
  Higher scores indicate more pain interference. Scores that are >= 55 (i.e., one half a SD above the normative mean) are considered clinically elevated.
Time Frame: Baseline (week 0), 4 week assessment, 8 week assessment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
Score on a scale
  Baseline | 64.3 (6.7) | 64.4 (7.2) | 60.5 (5.3) | 61.0 (4.59)
  4 Weeks | 64.4 (6.4) | 64.9 (7.2) | 59.4 (5.3) | 61.0 (5.9)
  8 Weeks | 64.0 (9.0) | 61.7 (7.6) | 56.6 (8.7) | 56.1 (9.1)

8. Primary Outcome: Participant Satisfaction
Description: Participants answered a Global Satisfaction question about their satisfaction with using the Rose application "Taking all things into account, how satisfied are you with using the Rose web application?" 4 - Very Satisfied 3 - Somewhat Satisfied 2 - Neutral
  1 - Somewhat Dissatisfied 0 - Very Dissatisfied
Time Frame: 4 Week, 8 Week timepoints
Population: The number of participants who expressed satisfaction will using the application was prespecified to be aggregated for all participants because the milestone for this feasibility variable was the overall rates of the satisfaction ratings for those who used the application at least once (i.e., participants in both conditions), collapsed across condition. We were not interested in, or anticipated, any between-group difference in this variable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Study 1 | Study 2
Number analyzed (Participants) | 50 | 50
Score on a scale | 2.8 (0.9) | 3.4 (0.9)

9. Secondary Outcome: PROMIS Anxiety Short Form 7a
Description: Domain assessed: Anxiety. Ratings are summed and converted to T scores (Mean = 50 and SD = 10 in the normative sample).
  Higher scores indicate more anxiety. Scores that are >= 55 (i.e., one half a SD above the normative mean) are considered clinically elevated.
Time Frame: Baseline (week 0), 4 week assessment, 8 week assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
T-score
  Baseline | 58.0 (10.5) | 55.5 (10.9) | 57.8 (4.8) | 54.0 (7.4)
  4 Weeks | 60.4 (11.3) | 59.2 (13.7) | 57.4 (6.7) | 54.8 (9.6)
  8 Weeks | 58.2 (11.3) | 57.0 (12.4) | 55.4 (8.0) | 54.1 (10.2)

10. Primary Outcome: System Usability Scale (SUS)
Description: Scale title: System Usability Scale. Minimum - Maximum range: 0 to 100. Higher scores indicate more usability (ease of use). There are no subscale scores for this measure.
Time Frame: 8 Week Timepoint
Population: The system usability scores for those who used the application at least once were prespecified to be aggregated for all participants because participants in both conditions had access to the application. The feasibility milestone was overall system usability score in participants in both conditions. The two groups had access the same application, and therefore we were not interested in, or anticipated, any between-group difference in this variable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Study 1: Summary measure for all participants in both the Treatment/Control groups for Study 1.
- Study 2: Summary measure for all participants in both the Treatment/Control groups for Study 2.
Arm/Group | Study 1 | Study 2
Number analyzed (Participants) | 50 | 50
Score on a scale | 80.33 (16.05) | 87.31 (12.72)

11. Secondary Outcome: Number of Participants Using Opioids
Description: Domain assessed: Opioid Use How assessed: Single item asking participants to indicate whether or not they currently using any opioid mediations.
  Unit of measure is the number and rate of participants who indicated that they are currently using at least one opioid medication.
Time Frame: Baseline (week 0), 4 week assessment, 8 week assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
Number analyzed (Participants) | 26 | 24 | 26 | 24
Participants | 10 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Enrollment until the 8 week follow up timepoint
Description: Adverse Events were systematically assessed by including the following question at all survey timepoints: "Have you experienced any negative side effects since our last contact as a result of the study (Yes/No)". IF YES: Please specify the negative side effects.
  Participants could also self-report Adverse Events when receiving a survey reminder phone call from a staff coordinator.
Arm/Group | Study 1: 8 Week Treatment | Study 1: 4 Week Waitlist | Study 2: 8 Week Treatment | Study 2: 4 Week Waitlist
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 1/26 | 0/24 | 0/26 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study 1: 8 Week Treatment (N=26) | Study 1: 4 Week Waitlist (N=24) | Study 2: 8 Week Treatment (N=26) | Study 2: 4 Week Waitlist (N=24)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 — AE was reported on the 4 week online self-report assessment and staff completed a follow up phone call with the participant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT06050083/Prot_SAP_000.pdf
  • Informed Consent Form: Study 1 consent form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT06050083/ICF_001.pdf
  • Informed Consent Form: Study 2 consent form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT06050083/ICF_002.pdf